CLINICAL TRIAL: NCT00328120
Title: An Open, Multicentre Phase I Clinical Study to Assess the Tolerability of Fulvestrant 500 mg in Postmenopausal Women With Hormone Receptor Positive Advanced or Recurrent Breast Cancer
Brief Title: Faslodex 500mg Multiple Dose Tolerability Study in BC Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6995C00004; 9238IL/0062
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Advanced Breast Cancer
Keywords: Advanced breast cancer; Faslodex
MeSH Terms: interventions — Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — 500 mg intramuscular injection
  Other Names: Faslodex; ZD9238

SUMMARY:
The primary objective of this study is to assess the tolerability of 500mg fulvestrant in postmenopausal women with hormone receptor positive, advanced or recurrent breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Postmenopausal woman who fulfils any one of the following criteria:
* Histological or cytological confirmation of breast cancer
* Estrogen receptor positive (ER+) or progesterone receptor positive (PgR+).

Exclusion Criteria:

* Having received any one of the following therapy for advanced or recurrent breast cancer
* 2 or more regimens of hormonal therapy or immunotherapy or 2 or more regimens of chemotherapy, etc

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04; Primary Completion 2006-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the tolerability of 500mg fulvestrant | assessed when all patients have been in the study for 6 months

SECONDARY OUTCOMES:
Pharmacokinetics | each visit
Time to progression | assessed when all patients have been in the study for 6 months
ORR | assessed when all patients have been in the study for 6 months
Clinical benefit rate | assessed when all patients have been in the study for 6 months
Time to response | assessed when all patients have been in the study for 6 months
duration of response and changes in serum tumour markers | assessed when all patients have been in the study for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Breast Cancer Established Brands Team Medical Science Director, MD, Study Director — AstraZeneca
Locations (5):
- Japan (5):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Nagoyata
  - Research Site, Osaka
  - Research Site, Tokyo